CLINICAL TRIAL: NCT00851175
Title: Is Augmentation of PORH by Rosuvastatin Adenosine-receptor Mediated?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: G. Rongen MD PhD, RUNMC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: rosucaff2
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-03

CONDITIONS: Atherosclerosis; Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — Rosuvastatin Calcium; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (No Intervention): forearm bloodflow after 2,3, and 5 minutes of forearm ischemia
- 2 (Active Comparator): forearm bloodflow after 2,3, and 5 minutes of forearm ischemia with concommitant administration of caffeine (90 ug/min/100ml forearm volume) into the brachial artery of the experimental (=non dominant) arm
  Interventions: Drug: caffeine
- 3 (Experimental): forearm bloodflow after 2,3, and 5 minutes of forearm ischemia after 7 days oral treatment with rosuvastatin 1dd 20mg
  Interventions: Drug: rosuvastatin
- 4 (Active Comparator): forearm bloodflow after 2,3, and 5 minutes of forearm ischemia after 7 days oral treatment with rosuvastatin 1dd 20mg with concommitant administration of caffeine (90 ug/min/100ml forearm volume) into the brachial artery of the experimental (=non dominant) arm
  Interventions: Drug: rosuvastatin; Drug: caffeine

INTERVENTIONS:
Drug: rosuvastatin — 7 day treatment with rosuvastatin 1dd 20mg
  Arms: 3; 4
Drug: caffeine — intra-arterial (brachial artery of non dominant arm) administration of caffeine(90 ug/min/100ml forearm volume)for approximately 60 minutes
  Arms: 2; 4

SUMMARY:
Rationale:

Statins form a class of drugs that is widely prescribed for hypercholesterolaemia, specifically to reduce the risk on atherosclerosis by lowering LDL-cholesterol. Next to the effect for which the drug was originally developed, it became obvious that statins have several other beneficial effects. Such pleiotropic effects include the activation of ecto-5'-nucleotidase which can increase endogenous adenosine production (by dephosphorylation adenosine monophosphate into adenosine) and subsequently cause vasodilation. A recent study of Meijer et al (not yet published) showed that rosuvastatin significantly augments vasodilation after a brief period of ischemia (post occlusive reactive hyperaemia). However, it is not yet verified whether this increase in post occlusive reactive hyperaemia is truly caused by a rise of extracellular adenosine and subsequent adenosine receptor stimulation. In this study, the mechanism by which rosuvastatin augments post occlusive reactive hyperaemia will be investigated by blocking adenosine receptors with caffeine, a competitive A1 and A2 adenosine receptor antagonist. Caffeine is a substance that can be safely used in normal concentrations to block the adenosine receptor.

Hypothesis:

The augmenting effect of rosuvastatin on PORH is caused by an increase of extracellular adenosine formation and this effect can be diminished by blocking the adenosine receptor using caffeine.

Objective:

To study the influence of caffeine on post occlusive reactive hyperaemia before and after 7 days treatment with rosuvastatin.

Study design:

Open label cross-over design Study population: Healthy volunteers, 18-50 years of age

Intervention:

Eight volunteers will receive a 7 day treatment with rosuvastatin 20 mg daily before and after rosuvastatin treatment caffeine will be administrated intra-arterially.

Main study parameters/endpoints:

Forearm blood flow (FBF) will be measured as an indicator for post occlusive reactive hyperaemia (PORH).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Written informed consent

Exclusion Criteria:

* History of any cardiovascular disease
* Hypertension (in supine position: systole >140 mmHg, diastole >90 mmHg)
* Diabetes Mellitus (fasting glucose >7.0 mmol/L or random glucose >11.0 mmol/L)
* Hyperlipidemia (fasting total cholesterol >5.5 mmol/L or random cholesterol >6.5 mmol/L)
* Alanine amino transferase >90 U/L
* Creatin kinase >440 U/L
* Raised rhabdomyolysis risk (GFR <80 ml/min and/or overt clinical signs of hypothyroidism and/or myopathy in family history
* Alcohol abuse
* Concommitant chronic use of medication
* Participation to any drug-investigation during the previous 60 days as checked with VIP check

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow (FBF)after 2, 5, and 13 minutes of forearm ischemia | before and after 7 day treament with rosuvastatin, with and without concommitant intra-arterial treatment with caffeine

CONTACTS AND LOCATIONS:
Overall Officials: G Rongen, MD PhD, Principal Investigator — RUNMC
Locations (1):
- RUNMC, Nijmegen, Netherlands

REFERENCES:
- [Background] Meijer P, Wouters CW, van den Broek PH, Scheffer GJ, Riksen NP, Smits P, Rongen GA. Dipyridamole enhances ischaemia-induced reactive hyperaemia by increased adenosine receptor stimulation. Br J Pharmacol. 2008 Mar;153(6):1169-76. doi: 10.1038/bjp.2008.10. Epub 2008 Feb 11. PMID 18264130
- [Background] Bijlstra PJ, den Arend JA, Lutterman JA, Russel FG, Thien T, Smits P. Blockade of vascular ATP-sensitive potassium channels reduces the vasodilator response to ischaemia in humans. Diabetologia. 1996 Dec;39(12):1562-8. doi: 10.1007/s001250050615. PMID 8960843